CLINICAL TRIAL: NCT00229827
Title: Optimal Timing for Repair of Left-to-Right Shunt Lesions
Brief Title: Optimal Timing for Repair of Left to Right Shunt Lesions
Status: Terminated | Type: Observational
Why Stopped: sufficient data was collected
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-092
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Ventricular Septal Defects; Persistent Common Atrioventricular Canal
Keywords: pediatric health; cardiac; pediatric population; congenital heart surgery; left to right shunt lesions; heart surgery; Atrioventricular canal defects
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Endocardial Cushion Defects

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine the optimal timing for repair of left-to-right shunt lesions such as ventricular septal defects and atrioventricular canals.

DETAILED DESCRIPTION:
In the past, children with left-to-right shunt lesions such as ventricular septal defects and atrioventricular canal defects were palliated with a pulmonary artery band. This prevented injury to the pulmonary vasculature while the child grew to a size where complete repair could be undertaken. With the improvements in surgical technique and critical care, there is a push to do a primary complete repair for these defects at younger and younger ages. These operations should be delayed as long as possible to allow for growth but not so long that there is unnecessary heart failure and medication requirements. The primary aim is to determine the optimal timing for repair of left-to-right shunt lesions such as ventricular septal defects and atrioventricular canals. The secondary aim is to define the criteria for failing medical anti-congestive heart failure therapy. This study will be conducted through a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the congenital surgery database
* Patients who have undergone repair of ventricular septal defects
* Patients who have undergone repair of atrioventricular canal defects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the congenital surgery database
  * Patients who have undergone repair of ventricular septal defects
  * Patients who have undergone repair of atrioventricular canal defects
Sampling Method: Non-Probability Sample
Enrollment: 200
Dates: Start 2005-05; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States